CLINICAL TRIAL: NCT07329530
Title: Characterisation of the Inflammatory, Metabolic, and Mitochondrial Profiles in the Context of Post-Intensive Care Muscle Dysfunction
Brief Title: Metabolic and Muscle Profile in ICU Survivors
Acronym: IM3SI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anne-Françoise Rousseau (Other)
Responsible Party: Sponsor-Investigator, Anne-Françoise Rousseau, Associate Professor, University of Liege
Organization: University of Liege (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IM3SI
Record Dates: First submitted 2025-12-12; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Critical Illness; Major Abdominal Surgeries
MeSH Terms: conditions — Critical Illness | interventions — Body Composition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICU patients (Experimental): Lab and clinical investigations to characterize the metabolic and muscle profile
  Interventions: Diagnostic Test: Inflammation markers; Diagnostic Test: Blood nucleosomes; Diagnostic Test: Erythrocyte membrane fatty acid content; Diagnostic Test: measurement of myokines; Diagnostic Test: Resting energy expendure; Diagnostic Test: body composition; Diagnostic Test: Omics; Diagnostic Test: Monocyte profile
- Surgical patients (Active Comparator): Lab and clinical investigations to characterize the metabolic and muscle profile
  Interventions: Diagnostic Test: Inflammation markers; Diagnostic Test: Blood nucleosomes; Diagnostic Test: Erythrocyte membrane fatty acid content; Diagnostic Test: measurement of myokines; Diagnostic Test: Resting energy expendure; Diagnostic Test: body composition; Diagnostic Test: Omics; Diagnostic Test: Monocyte profile

INTERVENTIONS:
Diagnostic Test: Inflammation markers — measurement of CRP, cytokines, MPO, oxidative stress during the first 7 days after ICU admission, between 1 and 7 days after ICU discharge and 3 months after ICU discharge (or the day after surgery and 3 months after hospital discharge)
Diagnostic Test: Blood nucleosomes — measurement of blood nucleosomes between 1 and 7 days after ICU discharge and 3 months after ICU discharge (or the day after surgery and 3 months after hospital discharge)
Diagnostic Test: Erythrocyte membrane fatty acid content — assessment of Erythrocyte membrane fatty acid content between 1 and 7 days after ICU discharge and 3 months after ICU discharge (or the day after surgery and 3 months after hospital discharge)
Diagnostic Test: measurement of myokines — measurement of myokines between 1 and 7 days after ICU discharge and 3 months after ICU discharge (or the day after surgery and 3 months after hospital discharge)
Diagnostic Test: Resting energy expendure — assessment of REE by indirect caloriometry during the first 7 days after ICU admission, between 1 and 7 days after ICU discharge and 3 months after ICU discharge (or the day after surgery and 3 months after hospital discharge)
Diagnostic Test: body composition — assessment of body composition by BIA during the first 7 days after ICU admission, between 1 and 7 days after ICU discharge and 3 months after ICU discharge (or the day after surgery and 3 months after hospital discharge)
Diagnostic Test: Omics — Blood metabolic, lipidomic, proteomic study during the first 7 days after ICU admission (or the day after surgery)
Diagnostic Test: Monocyte profile — Blood leukocyte and monocyte profiles and transcriptomic analysis between 1 and 7 days after ICU discharge and 3 months after ICU discharge (or the day after surgery and 3 months after hospital discharge)

SUMMARY:
More and more patients survive a critical illness requiring admission to the intensive care unit, but they may be left with sequelae that are independent of the initial pathology. From a physical standpoint, the most visible complication is intensive care unit-acquired muscle weakness. A major factor in the development and persistence of muscle dysfunction appears to be the inflammatory response and the neuroendocrine stress response triggered by the initial critical insult. Persistence of inflammation beyond ICU discharge has been demonstrated in several studies. In response to inflammation, there is also increased oxidative stress associated with mitochondrial dysfunction.

The objectives of the present study are therefore:

to determine whether the broad inflammatory and metabolic profile of patients who have survived an ICU stay can predict the trajectory of muscle performance over the three months following ICU discharge; to compare this profile and muscle performance with those of non-critically ill surgical patients who have undergone a standardized inflammatory stress of lower intensity than that associated with critical illness; to investigate mitochondrial function in skeletal striated muscle after ICU stay, in light of the inflammatory and metabolic profile; to assess whether abnormalities in mitochondrial function also affect tissues other than skeletal muscle, in particular circulating blood mononuclear cells.

ELIGIBILITY:
Inclusion Criteria

* Critical illness:
* anticipated ICU stay >= 7 days
* Major abdominal surgery
* elective surgery

Exclusion Criteria:

* Active malignancy
* Inherited metabolic disorder
* Known muscle disease
* Pregnancy
* Patient refusal
* Patient unable to express informed consent (dementia, confusion)
* Known coagulation disorder (cirrhosis, genetic coagulopathy) or thrombocytopenia < 100,000/mm³ on the day of biopsy, anemia with hemoglobin < 9 g/dL on the day of biopsy, or treatment with anticoagulant agents (contraindication to muscle biopsies only)
* Pacemaker or other implanted electronic device (contraindication to bioelectrical impedance analysis only)
* Oxygen therapy (contraindication to indirect calorimetry during spontaneous ventilation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Quadriceps strength | between 1 and 7 days after ICU discharge and 3 months after ICU discharge in the critically ill patients, or the day after the surgery and 3 months after the surgery in surgical patients
  Quadriceps strength in Newton, measured using a handheld dynamometer (MicroFet)
Handgrip strength | between 1 and 7 days after ICU discharge and 3 months after ICU discharge in the critically ill patients, or the day after the surgery and 3 months after the surgery in surgical patients
  Hangrip strength in kg, measured young an handheld dynamometer (Jamar)
Muscle mass | between 1 and 7 days after ICU discharge and 3 months after ICU discharge in the critically ill patients, or the day after the surgery and 3 months after the surgery in surgical patients
  Quadriceps muscle thickness assessed by ultrasound
Muscle mass | between 1 and 7 days after ICU discharge and 3 months after ICU discharge in the critically ill patients, or the day after the surgery and 3 months after the surgery in surgical patients
  Muscle mass assessed using bioelectrical impedance analysis
Muscle mitochondrial function | between 1 and 7 days after ICU discharge and 3 months after ICU discharge in the critically ill patients, or perioperatively and 3 months after the surgery in surgical patients
  Oxygraphy performed on a muscle sample
Muscle function | between 1 and 7 days after ICU discharge and 3 months after ICU discharge in the critically ill patients, or perioperatively and 3 months after the surgery in surgical patients
  Transcriptomic analysis in muscle sample (muscle biopsy)
Physical function | between 1 and 7 days after ICU discharge and 3 months after ICU discharge (or the day after surgery and 3 months after hospital discharge)
  2-minute walking test

OTHER OUTCOMES:
Health-related Quality of life | 3 months after ICU discharge in the critically ill patients, or 3 months after the surgery in surgical patients
  EQ-5D-3L questionnaire (3-level version of the EuroQOL questionnaire, including EQ-5D descriptive system with higher score indicating worst quality of life and the EQ visual analogue scale ranging from 0 to 100, with higher score indicating best quality of life)
Autonomy for ADL | 3 months after ICU discharge in the critically ill patients, or 3 months after the surgery in surgical patients
  Barthel index, ranging from 0 to 100, with higher score indicating full independency for activities of daily living
Health-related quality of life | 3 months after ICU discharge in the critically ill patients, or 3 months after the surgery in surgical patients
  SARQOL questionnaire (Sarcopenia and Quality Of Life questionnaire) - short form, ranging from 0 to 100, with higher score indicating best quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sart Tilman, Liège, Belgium